CLINICAL TRIAL: NCT00884182
Title: Safety and Immunogenicity of an Intramuscular A/H5N1 Inactivated, Split Virion Pandemic Influenza Vaccine in European Children
Brief Title: Safety and Immunogenicity of an Intramuscular A/H5N1 Inactivated, Split Virion Pandemic Influenza Vaccine in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GPA12
Record Dates: First submitted 2009-04-16; First posted 2009-04-20 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Influenza; Orthomyxoviridae Infections; Orthomyxovirus Infections
Keywords: Influenza; Orthomyxoviruses; Split Virion Pandemic Influenza Vaccine; A/H5N1
MeSH Terms: conditions — Influenza, Human; Orthomyxoviridae Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Experimental): Participants on vaccination schedule 1 (Day 0 and Day 21)
  Interventions: Biological: A/H5N1 Inactivated, Split Virion Pandemic Influenza Vaccine
- Group 2 (Experimental): Participants on vaccination schedule 2 (Day 0 and Day 14)
  Interventions: Biological: A/H5N1 Inactivated, Split Virion Pandemic Influenza Vaccine
- Group 3 (Experimental): Participants on vaccination schedule 3 (Day 0 and Day 42)
  Interventions: Biological: A/H5N1 Inactivated, Split Virion Pandemic Influenza Vaccine

INTERVENTIONS:
Biological: A/H5N1 Inactivated, Split Virion Pandemic Influenza Vaccine — 0.5 mL, Intramuscular

SUMMARY:
This study is part of an effort to develop an effective vaccination program in children in the event of a pandemic.

Study objectives:

* To describe the safety profiles in the periods following each vaccination in subjects receiving different vaccination schedule.
* To describe the immune response after each vaccination in subjects receiving study vaccine.

DETAILED DESCRIPTION:
Study participants will receive two administrations of the investigational vaccine at one of 3 vaccination schedules.

ELIGIBILITY:
Inclusion Criteria :

All Subjects

* Subject and parent(s)/legal representative able to attend all scheduled visits and to comply with all trial procedures.
* Completion of vaccination according to the national immunization schedule

Subjects Aged ≥ 2 Years to < 18 Years:

* Aged ≥ 2 years to < 18 years on the day of inclusion.
* Provision of Informed Consent Form signed by the subject's the parent(s)/legal representative (and by an independent witness if required by local regulations). In addition, provision of Assent Form signed by subjects aged 8 to 11 years, and of Informed Consent Form signed by subjects ≥ 12 years.
* For a female of child-bearing potential, avoid becoming pregnant (use of an effective method of contraception or abstinence) for at least 4 weeks prior to each vaccination, until at least 4 weeks after each vaccination.

Subjects Aged ≥ 6 Months to < 2 Years:

* Aged ≥ 6 months to < 2 years on the day of inclusion.
* Born at full term of pregnancy (≥ 37 weeks) with a birth weight ≥ 2.5 kg.
* Provision of Informed Consent Form signed by the parent(s) or other legal representative (and by an independent witness if required by local regulations).

Exclusion Criteria :

All subjects

* Participation in another clinical trial investigating a vaccine, drug, medical device, or a medical procedure in the 4 weeks preceding trial vaccination
* Planned participation in another clinical trial during the present trial period
* Known or suspected congenital or acquired immunodeficiency, immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months, or long-term systemic corticosteroids therapy
* Known systemic hypersensitivity to any of the vaccine components or history of a life-threatening reaction to the trial vaccine or to a vaccine containing any of the same substances
* Chronic illness, at a stage that could interfere with trial conduct or completion, in the opinion of the investigator
* Current alcohol abuse or drug addiction that may interfere with the subject's ability to comply with trial procedures
* Receipt of Blood or blood-derived products in the past 3 months, that might interfere with the assessment of immune response
* Receipt of any vaccine in the 4 weeks preceding trial vaccination
* Planned receipt of any vaccine in the 4 weeks following any trial vaccination
* (Known) Human Immunodeficiency Virus (HIV), Hepatitis B surface (HBs) antigen or Hepatitis C seropositivity
* Previous vaccination against avian influenza with either the trial vaccine or another vaccine
* Thrombocytopenia, bleeding disorder or anticoagulants in the 3 weeks preceding inclusion contraindicating IM vaccination
* Subjects deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized without his/her consent
* Received oral or injected antibiotic therapy within the 72 hours prior to any blood draw

Subjects Aged ≥2 Years to <18 Years:

* For a female of child-bearing potential, known pregnancy or positive urine pregnancy test
* Breast-feeding female
* Febrile illness (temperature ≥ 37.5 °C) or moderate or severe acute illness/infection on the day of vaccination, according to investigator judgment

Subjects Aged ≥ 6 Months to < 2 Years:

* History of seizures
* Febrile illness (temperature ≥ 38 °C) or moderate or severe acute illness/infection on the day of vaccination, according to investigator judgment.

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 350 (Actual)
Dates: Start 2009-04; Primary Completion 2010-03 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
To provide information concerning the safety of the Split Virion Pandemic Influenza vaccine. | 21 days post-vaccination and entire study

SECONDARY OUTCOMES:
To provide information concerning the immunogenicity of Split Virion Pandemic Influenza vaccine. | 21 days post-vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Sanofi Pasteur Inc.
Locations (10):
- Finland (10):
  - Espoo
  - Helsinki
  - Jarvenpaa
  - Kuopio
  - Lahti
  - Oulu
  - Pori
  - Tampere
  - Turku
  - Vantaa

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com